CLINICAL TRIAL: NCT06694649
Title: Effectiveness of Prehabilitation in Patients Undergoing Radical Cystectomy: a Retrospective Analysis
Brief Title: Better in Better Out Cystectomy.
Acronym: BIBOCYS-1
Status: Not yet recruiting | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Other Study IDs: Z-2024064
Record Dates: First submitted 2024-11-12; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (3):
- Independent aerobic exercise
- Primary care physiotherapy in own area
- Full internal prehabilitation program

SUMMARY:
The current gold standard for non-metastatic muscle-invasive bladder cancer or treatment-refractory high-risk non-muscle-invasive bladder cancer is radical cystectomy (RC). This procedure is associated with high rates of perioperative complications (30-65%) and mortality (1.5-10%). Patients who require radical cystectomy often present with multiple co-morbidities, a certain degree of frailty, functional deficits, and a high level of past or current tobacco use. According to the "better in, better out" principle, it is likely that by improving the physical, nutritional and psychological status, a reduction in morbidity and mortality will be observed.

The literature suggests that multimodal prehabilitation may reduce complications and improve functional recovery after major cancer surgery. Therefore, the prehabilitation programme used in this study includes exercise training, dietary advice, psychological support and smoking cessation advice. Prehabilitation has been offered to a selection of patients with increased risk for postoperative complications since 01/05/2023.

At ZOL Genk, patients receive preparation for RC in one of three ways, depending on a balancing exercise that considers the patient's complexity and frailty, functionality, mobility and other factors. Patient preference and place of residence are also taken into account in determining the most appropriate preparation pathway. 1. The patient is solely encouraged to increase his fitness level by means of independent aerobic exercise. 2. The patient receives a prescription for primary care physiotherapy in his own area. 3. The patient undergoes our full internal prehabilitation program. The primary objective of this study is to compare these three different groups in terms of mortality, ICU length of stay, length of hospital stay, complication rate, type of complications and readmission rate. Finally, patient adherence will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary bladder cancer (cTa-4N0-3M0) who underwent RARC.

Exclusion Criteria:

* Patients who needed a semi-urgent cystectomy.
* Patients with severe cognitive or psychiatric impairment.
* Patients with a contraindication to perform physical exercise training or a cardiopulmonary exercise test (CPET).
* Metastatic or non-primary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target group of this study are patients who have undergone robot-assisted radical cystectomy (RARC) for primary bladder cancer since 01/01/2021 and who have participated in one of the three preoperative prehabilitation programmes:
  1. The patient is solely encouraged to increase his fitness level by means of independent aerobic exercise.
  2. The patient receives a prescription for primary care physiotherapy in his own area.
  3. The patient undergoes our full internal prehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ICU length of stay | Until 90 days after RC
Mortality | Until 3 years after RC
Length of hospital stay | Until 90 days after RC
Complication rate | Until 90 days after RC
Type of complications | Until 90 days after RC
Readmission rate | Until 90 days after RC

IPD SHARING:
Plan to Share IPD: No